CLINICAL TRIAL: NCT02070887
Title: Inhibiting COMT in Parkinson's Disease A Monocenter, Observational, Rater-blinded Trial of Entacapone in Parkinson's Disease
Brief Title: Inhibiting COMT in Parkinson's Disease
Status: Withdrawn | Type: Observational
Sponsor: Christian Baumann (Other)
Responsible Party: Sponsor-Investigator, Christian Baumann, Professor dr. med., University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: KEK-ZH 2013-0276
Record Dates: First submitted 2014-02-18; First posted 2014-02-25 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Entacapone
- No Entacapone

SUMMARY:
The overall aim of this observational study is to investigate the impact of COMT inhibition on homocysteine metabolism, vascular physiology and correlates of neurodegeneration in PD patients with certain COMT genotype. It is designed to evaluate effect size of Hcy lowering to secondary outcome parameters. Assessment of outcome parameters will be rater-blinded or computer-based.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 - 75 years,
* Caucasian ethnicity,
* diagnosed PD by UK brain bank criteria,
* Hoehn & Yahr scale 2 - 3,
* fertile females have to use contraception
* Group 1: medication with Stalevo® (L-DOPA/DDI + Entacapone)
* Group 2: medication with Madopar® or Sinemet® (L-DOPA/DDI)

Exclusion Criteria:

* methotrexate therapy during the last 12 months,
* treatment with Tolcapone
* vitamin B6, B12 and/or folic acid supplementation during last 6 months,
* pregnancy,
* intention to become pregnant during the course of the study,
* breast feeding,
* other clinically relevant concomitant disease states by discretion of the investigator
* known or suspected non-compliance, drug or alcohol abuse,
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia or confusional state of the subject,
* participation in another study with investigational drug within the 30 days preceding and during the present study,
* enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary movement disorder clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Estimated); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Serum level of homocysteine | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christian Baumann, MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland